CLINICAL TRIAL: NCT03906903
Title: Effect of Transcranial Magnetic Stimulation as an Enhancer of a Cognitive Stimulation Maneuver in Mild Cognitive Impairment
Brief Title: Transcranial Magnetic Stimulation and Cognitive Stimulation in Mild Cognitive Impairment
Acronym: rTMS&MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Queretaro (Other)
Responsible Party: Principal Investigator, Dr. Julian Reyes López, Clinical Professor, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 05-01/02/2018
Record Dates: First submitted 2019-02-05; First posted 2019-04-08 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the clinical effects of 5Hz rTMS over Left Dorsolateral Prefrontal Cortex on an active versus placebo modality stimulation and Cognitive Stimulation.
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 Hz Stimulation (Active Comparator): This group will receive 5Hz (Hertz) Left Dorsolateral Prefrontal Cortex repetitive Transcranial Magnetic Stimulation with 1500 pulses per session, three per weekday, with a final result of 30 sessions in this modality with a 30 minutes Cognitive Stimulation after session.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Behavioral: Cognitive Stimulation
- Placebo Stimulation (Placebo Comparator): This group will receive the Sham modality simulating 1500 pulses of 5Hz Transcranial Magnetic Stimulation for 30 sessions, three per weekday with a 30 minutes Cognitive Stimulation afterwards.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Behavioral: Cognitive Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Subjects will receive both active and placebo rTMS, in a crossover modality.
  Other Names: Transcranial Magnetic Stimulation
Behavioral: Cognitive Stimulation — Subjects will receive 30 sessions of 30 minutes with Cognitive Stimulation in three areas (attention, memory and executive functions), one each week.

SUMMARY:
This study evaluates the effect of 5Hertz (Hz) repetitive Transcranial Magnetic Stimulation (rTMS) on Left Dorsolateral Prefrontal Cortex enhancing Cognitive Stimulation in Mild Cognitive Impairment.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is defined as an intermediate state between normal aging and an early stage of neurodegenerative diseases. It is estimated that exist 24.3 million people worldwide with neurocognitive disorders. Cognitive Stimulation (CS) is defined as the set of techniques and strategies that optimize the effectiveness in various functions of different cognitive abilities throughout its use in rehabilitation on MCI. Transcranial Magnetic Stimulation (rTMS) is a safe neuromodulation technique that modifies brain electrical activity through electromagnetic fields. There is evidence of the relationship between CS and rTMS for the improvement in MCI levels and cognitive functions; it´s important to deepen the knowledge of the therapeutic potential of both techniques combined on MCI

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both genders.
* Subjects from 60 to 85 years old.
* Meet Diagnostic and Statistical Manual, 5th edition (DSM-5) diagnostic criteria for Mild Cognitive Impairment.
* Patients must provide their oral and written informed consent.

Exclusion Criteria:

* Subjects with history of traumatic brain injury with loss of consciousness.
* Subjects with intracranial metallic objects or metal plates in the skull.
* Subjects diagnosed with uncontrolled chronic (for example: hypertension, diabetes) or neurological diseases.
* Comorbidity with other mental illness.
* Presence of psychotic symptoms, Bipolar Disorder and Substance abuse.
* Alterations in the electroencephalogram (epileptiform activity).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 24 weeks.
  MoCA is a test that evaluates the presence of Mild Cognitive Impairment.
Mini Mental State Examination (MMSE) | 24 weeks
  MMSE is a test that seeks the presence of Mild Cognitive Impairment
Attention and Memory Neuropsychological Battery (NEUROPSI) | 24 weeks
  NEUROPSI is a battery that evaluates the level of the Cognitive Impairment.

SECONDARY OUTCOMES:
Changes in Depressive symptoms evaluated by Geriatric Depression Scale (GDS - Yesavage - Brink) | 2 Weeks
  The Geriatric Depression Scale is a 30 item scale that evaluates the severity of depressive symptoms in Geriatric patients. With a minimum of 0 and a maximum of 30 scores, above 11 are suggestive for depression, relating a higher score with a higher depression level.
Changes in impulsive behavior evaluated by Barratt Impulsivity Scale (BIS-11) | 1 week
  The Barratt Impulsivity Scale is a likert-type self-questionnaire designed to assess the personality and behavioral construct of impulsiveness; composed of 30 items, each one scored from 0-4 according to the presence and severity of them, describing common impulsive or non-impulsive behaviors and preferences. This scale does not have a cut-off point, relating a higher score with a higher impulsivity in which can be assessed three types of impulsivity (cognitive, motor and non-planned impulsivity).

CONTACTS AND LOCATIONS:
Overall Officials: Julian V Reyes López, Psychiatrist, Study Director — Faculty of Medicine, Autonomous University of Queretaro
Locations (1):
- Autonomous University of Queretaro, Querétaro City, Querétaro, Mexico